CLINICAL TRIAL: NCT02304315
Title: A Randomized, Open-label, Single-center, Phase II Trial to Explore the Safety and Efficacy of GC1102 and Determine Its Optimal Dose After Intravenous Administration in HBV-related Liver Transplant Recipients
Brief Title: A Phase 2 Study of GC1102 (Recombinant Hepatitis B Immunoglobulin) in HBV-related Liver Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC1102_P2
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis B Infection
Keywords: HBV-related liver transplantation; Hepatitis B Immuno Globulin
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GC1102 50,000 IU (Experimental): Anhepatic phase: 50,000 IU intravenous during surgery, Post-transplantation(1st week): 50,000 IU intravenous every day, Post-transplantation(2nd-4th weeks): 50,000 IU intravenous every weeks, Post-transplantation(8th weeks and till 24 weeks): 50,000 IU intravenous every 4 weeks.
  Interventions: Biological: GC1102 50,000 IU
- GC1102 80,000 IU (Experimental): Anhepatic phase: 80,000 IU intravenous during surgery, Post-transplantation(1st week): 80,000 IU intravenous every day, Post-transplantation(2nd-4th weeks): 80,000 IU intravenous every weeks, Post-transplantation(8th weeks and till 24 weeks): 80,000 IU intravenous every 4 weeks.
  Interventions: Biological: GC1102 80,000 IU

INTERVENTIONS:
Biological: GC1102 50,000 IU — a recombinant hepatitis B immunoglobulin
  Arms: GC1102 50,000 IU
Biological: GC1102 80,000 IU — a recombinant hepatitis B immunoglobulin
  Arms: GC1102 80,000 IU

SUMMARY:
This is a proof-of-concept study for GC1102 to demonstrate preventing the recurrence of hepatitis B virus (HBV) infection following liver transplantation and a dose-finding study to determine its optional dose.

DETAILED DESCRIPTION:
GC1102 is a new recombinant hepatitis B immunoglobulin (HBIg) from Chinese Hamster Ovary (CHO) cells. It is a monoclonal antibody and has high affinity and avidity to hepatitis B surface antigen and several advantages compared to HBIg derived from blood plasma of human donors. Forty volunteers will participate in the study, receive 24-week treatment with low dose (50,000IU) of GC1102 or with high dose (80,000IU) and be followed up till 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Aged 19 - 65 years
* Expected liver transplantation related to hepatitis B
* Positive HBsAg

Exclusion Criteria:

* Patients has participated in any other clinical trial within 30 days
* Patients who are scheduled re-operation for liver transplantation
* Patients with are co-infected with HAV, HCV or HIV
* History of malignant tumor within 5 years except primary liver cancer
* Patients with moderate or severe renal disorder (serum creatinine > 1.5 X ULM) or anuria, acute renal failure or dialysis
* Patients who had experienced cardiovascular attack, myocardiac infarction, PTCA or coronary bypass or with angina, arrhythmia, or any other clinically meaningful valvular heart disease, cerebral infarction or cerebral hemorrhage within 6 months
* History of anaphylaxis against active ingredient or excipients of study drug
* Patients who had been vaccinated with parenteral live vaccine (measles vaccine, epidemic parotitis vaccine, rubella vaccine, cholera vaccine, chickenpox vaccine) within 3 months
* Patients who had been treated with any other immuno globulin within 3 months
* Pregnant or breast-feeding women
* Women of childbearing potential who do not agree to use appropriate contraceptive methods (condom, an intrauterine device, oral contraceptive hormones, or a vasectomy of male sex partner) during this study
* Alcohol or drug abuse within 6 months
* Patients who has any clinically meaningful disease in investigator's judgement to prevent participating in this study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of Hepatitis B | 28 weeks
  Seroconversion rate of HBsAg or HBeAg

SECONDARY OUTCOMES:
Seroconversion rate of HBsAg or HBeAg | 28 weeks
Seroconversion time of HBsAg or HBeAg | 28 weeks
Overall survival rate | 28 weeks
Geometric mean titer (GMT) of HBV DNA | Day 6, 28, 59, 84, 112, 140, 158, 196
Histological findings of hepatic graft | Baseline
  if available
Incidence rate of Anti-GC1102 Antibody | 28 weeks
Mutation rate of HBV DNA | 28 weeks

OTHER OUTCOMES:
Adverse events | 28 weeks
Clinical abnormalities in physical exam, vital signs, and/or laboratory | 28 weeks
Infusion reactions | 72 hours
  Any adverse events occurred within 72 hours after intervention
Pharmacokinetic parameters of GC1102 titer (C trough, t 1/2b, AUC, C max, and T max) | Day 6, 28, 59, 84, 112, 140, 158, 196
  C trough, t 1/2b, AUC, C max, and T max

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Gyu Lee, M.D., Principal Investigator — Seoul Asan Medical Center; Chang-Hee Lee, M.D., Study Director — GC Biopharma Corp
Locations (1):
- Seoul Asan Medical Center, Seoul, South Korea